CLINICAL TRIAL: NCT05149274
Title: A Randomized, Open-label Study to Evaluate the Pharmacokinetics and Safety of DWP14012 Tablet A and Compare Those of DWP14012 Tablet B in Healthy Subjects
Brief Title: Evaluate the Pharmacokinetics and Safety of DWP14012 Tablet A and Compare Those of DWP14012 Tablet B in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP14012107
Record Dates: First submitted 2021-11-15; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Phase 1 Study, Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part1 (Active Comparator): DWP14012 Tablet A : single/multiple dose, 1 group, 2 period study
  Interventions: Drug: DWP14012 Tablet A
- Part2 (Active Comparator): DWP14012 Tablet A 4T vs DWP14012 Tablet B 1T
  Interventions: Drug: DWP14012 Tablet A; Drug: DWP14012 Tablet B

INTERVENTIONS:
Drug: DWP14012 Tablet A — DWP14012 10mg
Drug: DWP14012 Tablet B — DWP14012 40mg
  Arms: Part2

SUMMARY:
The pharmacokinetics (PK) and safety of oral DWP14012 tablet A will be evaluated and compared with those of DWP14012 tablet B in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults >=19years and <=45 years of age
* BMI >=17.5 kg/m2 and <30.5kg/m2, and body weight >= 55kg for male and >= 45kg for femlae
* subjects with no abnormal symptoms or findings based on physical examinations
* subjects determined eligible based on the results of lab tests
* subjects who agree to participate

Exclusion Criteria:

* Subjects with medical history that can not be participated
* Subjects with results of lab tests performed at screening which meet any of the following :

  * ALT or AST > 1.5 times the upper limit of normal
  * Diagnosis of Helicobacter pylori (H. pylori) positive result
* subject who is allergic to IP
* subject with history of serious alcohol or drug abuse within 1 year prior to screening.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
(part 2) AUC last of DWP14012 | 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours after dosing
(part 2) Cmax of DWP14012 | 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours after dosing

SECONDARY OUTCOMES:
(Part 2) AUC inf of DWP14012 | 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours after dosing
(Part 2) Tmax of DWP14012 | 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours after dosing
(Part 2) t1/2 of DWP14012 | 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours after dosing
(part 1-period 1) AUC last of DWP14012 | 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours
(part 1-period 1) Cmax of DWP14012 | 0 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours
(part 1- period 2) AUC last of DWP14012 | 0 hours (pre-dose) on Day 5; 12 hours (pre-dose) on Day 7; 0 hours (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 (pre-dose), 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20, 24, and 48 hours after dosing on Day 8
(part 1- period 2) Cmax of DWP14012 | 0 hours (pre-dose) on Day 5; 12 hours (pre-dose) on Day 7; 0 hours (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 (pre-dose), 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20, 24, and 48 hours after dosing on Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea